CLINICAL TRIAL: NCT03352102
Title: Effects of Neuromuscular Electrical Stimulation of the Quadriceps and Diaphragm in Critically Ill Patients: a Pilot Study.
Brief Title: Electrical Stimulation of the Quadriceps and Diaphragm in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pericles Almeida Delfino Duarte (Other)
Responsible Party: Sponsor-Investigator, Pericles Almeida Delfino Duarte, MD, PhD, Universidade Estadual do Oeste do Paraná
Organization: Universidade Estadual do Oeste do Paraná (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134673
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Critical Illness Myopathy; Respiration, Artificial
Keywords: Electric Stimulation; Intensive Care Units; Mechanical Ventilation; Ventilator Weaning
MeSH Terms: conditions — Respiratory Aspiration | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diaphragm Group (DG) (Experimental): subjects who received conventional physical therapy once a day, plus a daily session of electrical stimulation in the diaphragm.
  Intervention: Electrical stimulation of the diaphragm.
  Interventions: Procedure: Electrical stimulation
- Quadriceps Group (QG) (Active Comparator): subjects who also received conventional physical therapy once a day, plus a daily session of electrical stimulation in the quadriceps.
  Intervention: Electrical stimulation of the quadriceps.
  Interventions: Procedure: Electrical stimulation
- Control Group (CG) (No Intervention): subjects who received regular treatment, i.e., conventional physical therapy, which included gross motor therapy and respiratory therapy twice a day every day, including weekend, during their stay in the ICU.

INTERVENTIONS:
Procedure: Electrical stimulation — Neuromuscular electrical stimulation therapy was performed
  Arms: Diaphragm Group (DG); Quadriceps Group (QG)

SUMMARY:
Subjects in MV will be included, divided into 3 groups: (a) Control Group (CG), (b) Stimulation of Quadriceps (Quadriceps Group - QG), (c) Stimulation of Diaphragm (Diaphragm Group - DG). The QG and DG patients will receive consecutive daily electrical stimulation sessions at specific points from the first day of randomization until ICU discharge. Respiratory and peripheral muscle strength, MV time, length of hospitalization and functional independence score (the Functional Status Score-ICU) will be recorded.

DETAILED DESCRIPTION:
Objective: Evaluate the effectiveness of the Neuro Muscular Electrical Stimulation therapy in quadriceps versus diaphragm subjects on mechanical ventilation (MV). Subjects in MV will be included, divided into 3 groups: (a) Control Group (CG), (b) Stimulation of Quadriceps (Quadriceps Group - QG), (c) Stimulation of Diaphragm (Diaphragm Group - DG). The QG and DG patients will receive consecutive daily electrical stimulation sessions at specific points from the first day of randomization until ICU discharge. Respiratory and peripheral muscle strength, MV time, length of hospitalization and functional independence score (the Functional Status Score-ICU) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or more
* 24 hours of MV or more

Exclusion Criteria:

Hemodynamic instability, pregnancy, body mass index(BMI) >35 kg/m2, history of neuromuscular disease at admission, brain death, diseases with systemic vascular involvement, bone fractures, use of an internal or external fixator, skin lesions, end-stage cancer, use of pacemakers, spinal injuries, or inability to receive an Medical Research Council score because of the cognitive state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
ICU and Hospital length of stay | 60 days
  Length of stay (in days) in ICU and in hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pericles Duarte, Principal Investigator — Hospital Universitário do Oeste do Parana, Universidade Estadual do Oeste do Parana.
Locations (1):
- Hospital Universitário do Oeste do Paraná, Cascavel, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No